CLINICAL TRIAL: NCT02498288
Title: Bioequivalence Study for an Isotretinoin Pharmaceutical Preparation - Capsules. Open, Crossover, Randomized, Single Dose, Three Treatments, Three Periods and Six Sequences With Meal (Breakfast) Study
Brief Title: A Study to Determine Bioequivalence of Isotretinoin in Healthy Male Subjects Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200115
Record Dates: First submitted 2013-05-16; First posted 2015-07-15 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
Keywords: capsule; Isotretinoin; Bioequivalence
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isotretinoin Arm (Experimental): All subjects in this study will be randomized to receive all the 3 distinct medications of isotretinoin in a sequential manner. Subjects will receive a single dosage of two capsules x 20 mg (40 mg) orally, for three periods, six sequences, with a wash-out period of two weeks to eliminate the first dosage.
  Interventions: Drug: Isotretinoin: Reference Medication 1; Drug: Isotretinoin: Reference Medication 2; Drug: Isotretinoin: Test Medication

INTERVENTIONS:
Drug: Isotretinoin: Reference Medication 1 — Isotretinoin reference medication 1 will be 40 mg in the pharmaceutical form of capsule (2 capsules of 20 mg each)
Drug: Isotretinoin: Reference Medication 2 — Isotretinoin reference medication 2 will be 40 mg in the pharmaceutical form of capsule (2 capsules of 20 mg each)
Drug: Isotretinoin: Test Medication — Isotretinoin test medication will contain isotretinoin 40 mg (2 capsules of 20 mg each) in the same type of pharmaceutical presentation, containing the same drug but possible to have a different excipients.

SUMMARY:
This is an open-label, crossover, randomized, single dose, three treatments, three periods and six sequences, single dosage, balanced study to determine Bioequivalence of Isotretinoin. Bioequivalence will be compared between the reference medication one (T1) vs the test medication (T3): (T1 vs T3); and the reference medication two (T2), vs test medication (T3): (T2 vs T3). Finally, treatments T1 vs T2 will be compared statistically to determine if they are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Included in study will be male volunteers.
* Ages between 18 and 45 years old.
* BMI (Body Mass Index) between 20 to 26 kilogram/meter square (kg/m^2).
* Anti-doping tests negative results.
* Negative test results for Ac human immunodeficiency virus (HIV), HBsAg (hepatitis B surface antigen), and rapid plasma regain (RPR; syphilis test).
* Clinical biochemical test values: Hematic Biometry, Urine Analysis, Biochemical Profile: (Glucose, Ureic Nitrogen, Urea, Creatinine, Uric Acid, Cholesterol, Triglycerides, Total Proteins, Albumin, Globulin, Bilirubin (total, indirect and direct), Alkaline Phosphatase (ALP), Lactic Dehydrogenase, Asparate aminotransferase (AST), Alanine aminotransferase (ALT), Calcium, Phosphorus, Sodium, Potassium, Chlorine and Iron), Ac HIV, HBsAg and RPR, must fall within an interval between minimum and maximum values in connection to said tests accepted values.
* Normal Electrocardiogram (ECG) and Chest X-rays.
* Complete the scale 'Columbia Suicide Severity Rating Scale' (C-SSRS), before and after each dosification period.
* Obtain a grade of zero in the C-SSRS.
* Signed the Informed Consent corresponding to the bioequivalence study.
* In exception cases, accepted may be a candidate for which any previously mentioned test is exceeded regarding considered valid maximum and minimum accepted normal values, as long as it involves an isolated value and there are no other manifestations which could allow assuming that a given value is related to a disease or is remnant of another. These cases must be approved by clinical area and declared as "Non-clinically significant".

Exclusion Criteria:

* Electrocardiographic Anomalies; radiological
* Anti-doping tests positive results,
* Positive results regarding RPR; HIV and HBsAg tests.
* Personal or family history of allergy to medication in question.
* Having any kind of allergy, since these persons are in higher risk of suffering from medication allergy.
* Tobacco use.
* Persons undergoing any medical treatment.
* Existence of concurrent or intercurrent disease.
* History psychiatric disorder (eg, Major Depressive Disorder, Generalized Anxiety Disorder, Bipolar Disorder (I or II), or schizophrenia).
* Existence of justified doubt regarding questionnaire answers truthfulness.
* Having participated in bioequivalence or bioavailability studies or having donated blood 2 months before the study.
* Presence of clinically important gastrointestinal diseases or malabsorption history during the last year.
* Presence of a medical condition requiring regular medication (with prescription or over-the- counter medication) with systemic absorption.
* Drugs or alcohol addiction history requiring treatment.
* Refuse to take the scale 'C-SSRS, before and after each dosification period.
* Obtain a grade greater than zero in the C-SSRS.
* Do not sign the Informed Consent corresponding to the bioequivalence study.
* Finally, excluded will be all those volunteers not meeting that established in Mexican Official Standard NOM-177-SSA1-1998.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2013-07-15 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero hours to last quantifiable time (AUC0-t) | Pre-dose and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours post dose in each treatment period
  Bioequivalence will be evaluated for isotretinoin 40 mg using three distinct medications; two assigned as reference medication (T1 and T2) and 1 test medication (T3). Each subject will receive 2 capsules (20 mg each) orally.
Area under the plasma concentration-time curve from zero hours to infinite (AUC0-infinity) | Pre-dose and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours post dose in each treatment period
  Bioequivalence will be evaluated for isotretinoin 40 mg using three distinct medications; two assigned as reference medication (T1 and T2) and 1 test medication (T3). Each subject will receive 2 capsules (20 mg each) orally.
Maximum drug concentration (Cmax) | Pre-dose and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours post dose in each treatment period
  Bioequivalence will be evaluated for isotretinoin 40 mg using three distinct medications; two assigned as reference medication (T1 and T2) and 1 test medication (T3). Each subject will receive 2 capsules (20 mg each) orally.
Time to maximum drug concentration (Tmax) | Pre-dose and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours post dose in each treatment period
  Bioequivalence will be evaluated for isotretinoin 40 mg using three distinct medications; two assigned as reference medication (T1 and T2) and 1 test medication (T3). Each subject will receive 2 capsules (20 mg each) orally.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Monterrey, Nuevo León, Mexico

REFERENCES:
- See also: Results for study 200115 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200115?search=study&study_ids=200115#rs